CLINICAL TRIAL: NCT02733796
Title: Persistence of Zika Virus in Semen After Acute Infection
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: B300201628191
Record Dates: First submitted 2016-03-30; First posted 2016-04-12 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Zika Virus; Zika Virus Disease; Virus Shedding; Transmission
Keywords: zika virus; semen analysis; sexual transmission
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sera urine semen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective observational laboratory evaluation of the persistence rate of zika virus (ZIKV) infection in semen by real-time Reverse Transcriptase Polymerase Chain Reaction (RT-PCR), and assessment of ZIKV replication-competence in semen by isolation of ZIKV. Evaluation of the persistence of ZIKV and its replication-competence in semen samples will increase the understanding of the risk of sexual transmission of ZIKV infection in the post-viremic phase in non-epidemic settings.

DETAILED DESCRIPTION:
Objectives

1. To assess the duration of persistence of zika virus (ZIKV) in semen samples by means of RT-PCR, after acute ZIKV infection.
2. To assess replication fitness of ZIKV in semen, by isolation of ZIKV virions in culture.

Study design, population, materials and methods: Prospective cohort study of persistence of zika virus (ZIKV) in semen samples of adult male patients who attend the outpatient clinic of the Institute of Tropical Medicine in Antwerp and who have a confirmed ZIKV infection (positive RT-PCR for ZIKV in a serum or urine sample at the time of inclusion). Clinical and epidemiological data will be recorded in a standardized Case Record Form (CRF). Baseline serum, blood and urine samples will be collected as required for routine clinical evaluation of an individual case and for arbovirus antibody detection assays; sampling of serum and urine collection for RT-PCR will be scheduled weekly until 2 consecutive semen samples test negative in ZIKV RT-PCR. ZIKV isolation will be attempted from each available semen sample with a positive PCR result. The semen analyses will include: sperm count, morphology, motility, leukocyte and erythrocyte count and pH of the semen. Serum at 4 weeks will be collected for ZIKV antibody detection assay.

Sample size : panel of 20 ZIKV confirmed cases Endpoints: Proportion of ZIKV positive RT-PCR on semen samples over time after confirmation of acute ZIKV infection, positivity rates of ZIKV isolation from semen samples over time after acute ZIKV infection.

Expected results and relevance : Evaluation of the persistence of ZIKV and its replication-competence in semen samples will increase the understanding of the risk of sexual transmission of ZIKV infection in the post-viremic phase in non-epidemic settings. This evidence will contribute to a more rational advice on preventing sexual transmission of ZIKV infection.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18 years or older
* Confirmed ZIKV case, defined as:

  * Having traveled to an affected area and developing at least 2 of the following Zika virus disease compatible symptoms within 2 weeks of travel: fever defined as T≥ 37.8°C (axillary measurement), maculopapular rash, arthralgia or non-purulent conjunctivitis.
  * Zika virus diagnosis by:RNA detection by RT-PCR in serum or urine during the first 10 days after infection, OR Four-fold or greater change in virus-specific quantitative antibody titers in paired sera, OR Virus-specific Immunoglobulin M (IgM) antibodies in serum with confirmatory virus-specific neutralizing antibodies in the same or a later specimen

Exclusion Criteria:

* History of, or ongoing urologic malignancy or urologic surgical treatment (including vasectomy).
* Recent (< 2 years) history of, or ongoing urinary tract infection (including prostatitis, epididymitis, sexually transmitted diseases).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men of 18 years or older, with confirmed ZIKV infection, residing in areas without epidemiologically important arthropod-borne ZIKV transmission
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of ZIKV persistence in semen | weekly followup (until 2 consecutive negative PCR results)- up to 6 months
  proportion of ZIKV positive semen samples in adult male patients after acute ZIKV infection over time

SECONDARY OUTCOMES:
kinetics of ZIKV persistence in semen | weekly followup (until 2 consecutive negative PCR results)- up to 6 months
  kinetics of ZIKV in semen samples by means of RT-PCR Cycle threshold (Ct-value) results after acute ZIKV infection over time
replication fitness of ZIKV in semen | weekly followup (until 2 consecutive negative PCR results)- up to 6 months
  assess replication fitness of ZIKV in semen, by isolation
comparison of ZIKV sequences from semen vs. non-semen samples | weekly followup (until 2 consecutive negative PCR results)- up to 6 months
  comparison of ZIKV sequences of virus isolated from semen vs. non-semen samples to detect potential compartmentalization

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bottieau, MD PhD, Study Chair — Institute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- ITM, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Yes, de-identified individual participant data will be made available for all primary and secondary study outcomes within 6 months of study completion
Time Frame: within 6 months of study completion
Access Criteria: Eligible researchers will be able to request access through a access request form

REFERENCES:
- [Background] Foy BD, Kobylinski KC, Chilson Foy JL, Blitvich BJ, Travassos da Rosa A, Haddow AD, Lanciotti RS, Tesh RB. Probable non-vector-borne transmission of Zika virus, Colorado, USA. Emerg Infect Dis. 2011 May;17(5):880-2. doi: 10.3201/eid1705.101939. PMID 21529401
- [Background] Musso D, Roche C, Robin E, Nhan T, Teissier A, Cao-Lormeau VM. Potential sexual transmission of Zika virus. Emerg Infect Dis. 2015 Feb;21(2):359-61. doi: 10.3201/eid2102.141363. PMID 25625872
- [Background] Gourinat AC, O'Connor O, Calvez E, Goarant C, Dupont-Rouzeyrol M. Detection of Zika virus in urine. Emerg Infect Dis. 2015 Jan;21(1):84-6. doi: 10.3201/eid2101.140894. PMID 25530324
- [Background] Hirayama T, Mizuno Y, Takeshita N, Kotaki A, Tajima S, Omatsu T, Sano K, Kurane I, Takasaki T. Detection of dengue virus genome in urine by real-time reverse transcriptase PCR: a laboratory diagnostic method useful after disappearance of the genome in serum. J Clin Microbiol. 2012 Jun;50(6):2047-52. doi: 10.1128/JCM.06557-11. Epub 2012 Mar 21. PMID 22442323
- [Background] Poloni TR, Oliveira AS, Alfonso HL, Galvao LR, Amarilla AA, Poloni DF, Figueiredo LT, Aquino VH. Detection of dengue virus in saliva and urine by real time RT-PCR. Virol J. 2010 Jan 27;7:22. doi: 10.1186/1743-422X-7-22. PMID 20105295
- [Background] Korhonen EM, Huhtamo E, Virtala AM, Kantele A, Vapalahti O. Approach to non-invasive sampling in dengue diagnostics: exploring virus and NS1 antigen detection in saliva and urine of travelers with dengue. J Clin Virol. 2014 Nov;61(3):353-8. doi: 10.1016/j.jcv.2014.08.021. Epub 2014 Sep 1. PMID 25242312
- [Background] Barzon L, Pacenti M, Franchin E, Pagni S, Martello T, Cattai M, Cusinato R, Palu G. Excretion of West Nile virus in urine during acute infection. J Infect Dis. 2013 Oct 1;208(7):1086-92. doi: 10.1093/infdis/jit290. Epub 2013 Jul 2. PMID 23821721
- [Background] Oster AM, Brooks JT, Stryker JE, Kachur RE, Mead P, Pesik NT, Petersen LR. Interim Guidelines for Prevention of Sexual Transmission of Zika Virus - United States, 2016. MMWR Morb Mortal Wkly Rep. 2016 Feb 12;65(5):120-1. doi: 10.15585/mmwr.mm6505e1. PMID 26866485
- See also: World Health Organization declares Public Health Emergency of International Concern — http://www.who.int/mediacentre/news/statements/2016/1st-emergency-committee-zika/en/